CLINICAL TRIAL: NCT00761449
Title: A Multicentre Phase II Study of the Efficacy and Safety of Lenalidomide in High-risk Myeloid Disease (High-risk MDS and AML) With a Karyotype Including Del(5q) or Monosomy 5
Brief Title: Lenalidomide in High-risk MDS and AML With Del(5q) or Monosomy 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic MDS Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMDSG07A; EudraCT no: 2007-000450-31
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2010-01

CONDITIONS: MDS; AML
Keywords: MDS; AML; Lenalidomide; monosomy 5; del5q
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 1. lenalidomide
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Initial dose is oral lenalidomide 10 mg daily continuously. The dose should be increased to 20 mg day 1 in week 6 and to 30 mg day 1 in week 10. This dose should be kept for seven weeks. Thus, the total study period is 16 weeks.
  Other Names: Revlimid

SUMMARY:
The aim of this study is to investigate the efficacy of lenalidomide in high risk MDS or AML with chromosome 5 aberrations.

DETAILED DESCRIPTION:
Previous studies have shown that the immunomodulatory drug lenalidomide is effective in the treatment of low risk MDS with del(5q). Treatment of this subgroup of MDS patients resulted in 67% major erythroid responses and 45% complete cytogenetic responses. We therefore intend to test the efficacy of lenalidomide in a group of high-risk patients who are ineligible for conventional chemotherapy and who have a dismal prognosis. The patients must have a karyotype including del(5q) but patients with a karyotype including monosomy 5 are also eligible. We hypothesize that hight risk MDS or AML patients with other chromosomal aberrations than del(5q) can be affected by the lenalidomide effect.

ELIGIBILITY:
Inclusion Criteria:

* Must be >18 years of age at the time of signing the informed consent form
* MDS at IPSS Int-2 or High with a karyotype including del(5q) or monosomy 5 confirmed with FISH (using the LSI EGR1/D5S23,D5S721 FISH probe)
* Acute myeloid leukemia with a karyotype including del(5q) or monosomy 5 confirmed with FISH (using the LSI EGR1/D5S23,D5S721 FISH probe)
* Patients could be included if:
* At diagnosis and not considered eligible for induction chemotherapy
* Refractory to induction therapy
* Relapse after induction chemotherapy leading to CR and considered not eligible for reinduction
* Relapse after allogeneic stem cell transplantation and not considered suitable for reinduction chemotherapy or other conventional relapse therapy.
* Subject has signed the informed consent document.
* Women of childbearing potential, WCBP, must agree to practice complete abstinence from heterosexual intercourse or to use two methods of contraception beginning 4 weeks prior to the start of the study medication, while on study medication and 4 weeks after the last dose of study medication. WCBP must have two negative serum or urine pregnancy tests prior to starting study drug. WCBP must agree to have pregnancy tests weekly for the first 4 weeks and then every 4 weeks while on study medication and 4 weeks after the last dose of study medication.
* Males (including those who have had a vasectomy) must use barrier contraception (latex condoms) when engaging in reproductive sexual activity with WCBP while on study medication and 4 weeks after the last dose of study medication.

Exclusion Criteria:

* Pregnant or lactating females.
* Prior therapy with lenalidomide
* Patients who are eligible for curative treatment
* Expected survival less than two months.
* Acute promyelocytic leukemia (APL)
* Absolute peripheral blast count >30,000/mm3
* Central nervous system leukemia
* Serum biochemical values as follows
* Serum creatinine >2.0 mg/dL (177 micromol/L)
* Serum aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) >3.0 x upper limit of normal (ULN)
* Serum total bilirubin >1.5 mg/dL (26 micromol/L)
* Prior allergic reaction to thalidomide
* Uncontrolled systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Major cytogenetic response (50% or more reduction of the del5(q) or monosomy 5 FISH positive clone in the bone marrow using the LSI EGR1/D5S23,D5S721 FISH probe) after 16 weeks of lenalidomide treatment | 16 weeks

SECONDARY OUTCOMES:
Minor and complete cytogenetic (FISH) response after 8 and 16 weeks | 16 weeks
Red blood cell transfusion independence | 16 weeks
Erythroid response | 16 weeks
Bone marrow response (morphology) | 16 weeks
Modification of gene expression profiling during treatment | 16 weeks
Safety | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hellström-Lindberg, MD, PhD, Principal Investigator — Nordic MDS Group
Locations (18):
- Denmark (6):
  - Department of Hematology, Aalborg Hospital, Aalborg
  - Department of Hematology, Aarhus University Hospital, Aarhus
  - Department of Hematology, Rigshospitalet, Copenhagen
  - Department of Hematology, Herlev Hospital, Herlev
  - Department of Hematology, Odense University Hospital, Odense
  - Department of Hematology, Vejle Hospital, Vejle
- Norway (3):
  - Department of Hematology, Rikshospitalet University Hospital, Oslo
  - Department of Medicine, Ullevål Hospital, Oslo
  - Department of Hematology, Trondheim University Hospital, Trondheim
- Sweden (9):
  - Department of Hematology and Coagulation, Sahlgrenska University hospital, Gothenburg
  - Department of Hematology, Lund University Hospital, Lund
  - Department of Hematology, Malmö University Hospital, Malmo
  - Department of Medicine, Örebro University Hospital, Örebro
  - Hematology Center, Karolinska University Hospital Huddinge, Stockholm
  - Hematology Center, Karolinska University Hospital Solna, Stockholm
  - Department of Medicine, Sundsvall Hospital, Sundsvall
  - Department of Medicine, Umeå University Hospital, Umeå
  - Department of Hematology, Akademiska University Hospital, Uppsala

REFERENCES:
- [Derived] Mollgard L, Saft L, Treppendahl MB, Dybedal I, Norgaard JM, Astermark J, Ejerblad E, Garelius H, Dufva IH, Jansson M, Jadersten M, Kjeldsen L, Linder O, Nilsson L, Vestergaard H, Porwit A, Gronbaek K, Hellstrom-Lindberg E. Clinical effect of increasing doses of lenalidomide in high-risk myelodysplastic syndrome and acute myeloid leukemia with chromosome 5 abnormalities. Haematologica. 2011 Jul;96(7):963-71. doi: 10.3324/haematol.2010.039669. PMID 21719884
- See also: Nordic MDS Group website — http://www.nmds.org